CLINICAL TRIAL: NCT02877212
Title: Association of FC Gamma RIIIA Polymorphism and Thrombopoietin (THPO) Expression With Response to TPO Agonists in Refractory ITP and the Impact of Therapy on B and T Cells Subsets in the Patients With Mutated Genotypes
Brief Title: Association of FcγRIIIA Polymorphism and THPO Expression With Response to Eltrombopag in Refractory ITP Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Parvez Ahmed, FCPS, MCPS, National Institute of Blood and Marrow Transplant (NIBMT), Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFBMTC_ITP_2016
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Immune Thrombocytopenic Purpura (ITP)
Keywords: ITP; Eltrombopag; Steroid refractory; Fc Receptor
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study subjects (Experimental): Steroid refractory ITP patients will be given Eltrombopag to investigate the association of treatment outcome with Fc Receptor polymorphism and THPO expression in responders and non responders following comparison correlation with ITP patients treated with standard IST as control group
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be given to steroid refractory ITP patients and ITP patients treated with standard Immunosuppressive therapy (IST) will be taken as control.
  Other Names: TPO Receptor agonists

SUMMARY:
Idiopathic thrombocytopenic purpura (ITP) is an autoimmune disease characterized by antibody-mediated platelet destruction. The complex pathogenesis of ITP with multiple challenges to immune system in terms of genetic predisposition, infection, responsiveness to immunosuppressive therapy (IST) and inhibition of platelet production has proven the diversity of constraints in diagnosing and treating ITP. Thrombopoietin receptor agonist (Eltrombopag) is specifically indicated for the treatment of thrombocytopenia in patients with chronic immune (idiopathic) thrombocytopenic purpura (ITP) who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy. This clinical trial aims to investigate the association of Fc gammaRIIIA gene (V158F) genetic predisposition with treatment outcome of Immune Thrombocytopenia (ITP) in refractory ITP patients and especially with Eltrombopag.

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura (ITP) is a autoimmune disorder in which a decreased number of circulating platelets (thrombocytopenia) manifests as a bleeding tendency, easy bruising (purpura), or extravasation of blood from capillaries into skin and mucous membranes (petechiae).

In persons with ITP, platelets are coated with autoantibodies to platelet membrane antigens, resulting in splenic sequestration and phagocytosis by mononuclear macrophages. The resulting shortened life span of platelets in the circulation, together with incomplete compensation by increased platelet production by bone marrow megakaryocytes, results in a decreased platelet count.

In immune thrombocytopenic purpura (ITP), an abnormal autoantibody, usually immunoglobulin G (IgG) with specificity for one or more platelet membrane glycoproteins (GPs), binds to circulating platelet membranes to induce clinically significant platelet dysfunction by directly blocking access of agonists to platelet Gp receptors.

Autoantibody-coated platelets induce Fc receptor-mediated phagocytosis by mononuclear macrophages, primarily but not exclusively in the spleen. The spleen is the key organ in the pathophysiology of ITP, not only because platelet autoantibodies are formed in the white pulp, but also because mononuclear macrophages in the red pulp destroy immunoglobulin-coated platelets.

Polymorphisms in FcγRIIIA have been implicated in responsiveness to splenectomy, corticosteroids and rituximab. Current trial is designed to investigate the impact of genetic predisposition of FcγRIIIA polymorphisms in refractory ITP patients treated with Eltrombopag along with cytokine profile expression in responders and non responders.

Eltrombopag is a small molecule thrombopoietin receptor agonist for oral administration. Eltrombopag interacts with the transmembrane domain of the thrombopoietin receptor (also known as cMpl) leading to increased platelet production.It is specifically indicated for the treatment of thrombocytopenia in patients with chronic immune (idiopathic) thrombocytopenic purpura (ITP) who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy.

Eltrombopag is supplied as a tablet designed for oral administration. In Pakistan, where patients; who are of East Asian ancestry or who have moderate to severe hepatic impairment, the recommended initial dose of Eltrombopag is 25 mg once daily. Eltrombopag should be adjusted to achieve and maintain a platelet count >50 x 109/L as necessary to reduce the risk for bleeding. The dosing of Eltrombopag should not exceed 75 mg daily.

Methodology:

1. Blood samples (serum, plasma, DNA*) will be collected from 50 controls (treated with standard immunosuppressive therapy (IST) as first and second line treatment) and 25 patients (steroids refractory) at the time of enrollment to the trial (pre-treatment; 0) and then sequentially at 3 and 6 months after treatment.
2. When a marrow analysis is indicated, some marrow specimens will also be collected and studied and if a patient to undergoes splenectomy as part of treatment, spleen specimens will also be collected and cryopreserved.
3. Fc gamma RIIIA V158F polymorphism will be assessed by means of an allele-specific PCR and/nested PCR following sequence verification
4. In order to validate the genotypes of study participants; direct sequencing of the SNPs will be done through automated capillary sequencing method.
5. Thrombopoietin (THPO) expression will be quantified before treatment and at 0, 3 and 6 months after treatment by real time PCR using house keeping gene (Beta Actin) as positive control in the refractory and control subjects.
6. The sequential analysis of T cells and anti-platelets (anti-GpIIbIIIa) antibodies producing B cells will be performed before and after treatment by means of flow cytometry in order to characterize T cells (TH1, TH2, TH17, TFH, Tregs subsets) and B cells (CD19+ representing B cell regulators).
7. Immune cells expressing cytokines in subjects with wild type and mutated genotypes will be measured to investigate its correlation with platelet recovery in responders and non responders by using Human Thrombopoietin Luminex performance Assay (R&D system Inc.; Bead-based multiplex assay for the Luminex® platform).
8. To find the association of the Fc V158F genotypic distribution with THPO and cytokine expression in THPO agonists responders and nonresponders ; statistical analysis will be performed by using statistical program SPSS (Version 23.0) .

ELIGIBILITY:
Inclusion Criteria:

* Steroid refractory ITP defined according to the recent consensual criteria (Rodeghiero F et al. Blood 2009),
* Informed consent. The control patients will be included as under;
* Age and sex matched controls
* Control ITP group (treated with standard immunosuppressive therapy (IST) as first and second line treatment)

Exclusion Criteria:

* Secondary ITP
* Other hematological and malignant disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The overall response rate 4-6 months after treatment defined by a platelet count > 30 x 109/L with at least a two-fold increase from the initial (pre-treatment) count | 6 months after inclusion
Fc Receptor polymorphism and THPO expression in responders and non-responders | 6-12 months after inclusion
  The inclusion of 75 patients (25 ITP patients treated with Eltrombopag and 50 subjects with ITP treated with other standard IST) would be considered as sufficient to show an association of the FcgammaRIIIA V158F genotypes distribution and THPO expression with the response for the patients treated with Eltrombopag and other IST at different time points; (M0, M3 and M6 )** **M0=pretreatment sample at 0 month; M3=sample after 3 months of treatment; M6= sample after 6 months of treatment.

SECONDARY OUTCOMES:
The Thrombopoietin and cytokine expression among the responders and non responders | 6 months
  The Thrombopoietin and cytokine expression among the responders and non responders will be taken as secondary outcome to evaluate the influence of Fc gamma RIIIA mutated genotypes to evaluate the correlation between steroid refractory and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Ahmed, FCPS, MCPS, Principal Investigator — Armed Forces Bone Marrow Transplant Centre, Rawalpindi, Pakistan; Andleeb Hanif, M.Phil, Study Director — andleebhanif123@gmail.com
Locations (1):
- Armed Forces Bone Marrow Transplant Centre, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erickson-Miller CL, Delorme E, Tian SS, Hopson CB, Landis AJ, Valoret EI, Sellers TS, Rosen J, Miller SG, Luengo JI, Duffy KJ, Jenkins JM. Preclinical activity of eltrombopag (SB-497115), an oral, nonpeptide thrombopoietin receptor agonist. Stem Cells. 2009 Feb;27(2):424-30. doi: 10.1634/stemcells.2008-0366. PMID 19038790
- [Background] Nimmerjahn F. Immunomodulation of immunothrombocytopenia. Semin Hematol. 2016 Apr;53 Suppl 1:S10-2. doi: 10.1053/j.seminhematol.2016.04.004. Epub 2016 Apr 6. PMID 27312154
- [Background] Akyol Erikci A, Karagoz B, Bilgi O. Regulatory T Cells in Patients with Idiopathic Thrombocytopenic Purpura. Turk J Haematol. 2016 Jun 5;33(2):153-5. doi: 10.4274/tjh.2015.0335. PMID 27211045
- [Background] Milosevic I, Slade E, Drysdale H; COMPare project team. Eltrombopag for chronic immune thrombocytopenia. Lancet. 2016 Jan 23;387(10016):336. doi: 10.1016/S0140-6736(16)00107-0. No abstract available. PMID 26842445